CLINICAL TRIAL: NCT00578682
Title: A Phase I, Randomized, Double-Blind, Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI-557, A Humanized Monoclonal Antibody With an Extended Half-Life Against Respiratory Syncytial Virus (RSV), in Healthy Adults
Brief Title: A Phase I, Randomized, Double-Blind, Single-Dose, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI-557
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: M. Pamela Griffin, M.D., MedImmune
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP144
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
MeSH Terms: interventions — motavizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): Single IV dose of 0.3 mg/kg MEDI-557
  Interventions: Biological: MEDI-557
- 2 (Experimental): Single IV dose of 3 mg/kg MEDI-557
  Interventions: Biological: MEDI-557
- 3 (Experimental): Single IV dose of 15 mg/kg MEDI-557
  Interventions: Biological: MEDI-557
- 4 (Experimental): Single IV dose of 30 mg/kg MEDI-557
  Interventions: Biological: MEDI-557

INTERVENTIONS:
Biological: MEDI-557 — Single IV dose of 3 mg/kg
  Other Names: motavizumab
  Arms: 2
Biological: MEDI-557 — Single IV dose of 15 mg/kg
  Other Names: motavizumab
  Arms: 3
Biological: MEDI-557 — Single IV dose of 30 mg/kg
  Other Names: motavizumab
  Arms: 4
Biological: MEDI-557 — Single IV dose of 0.3 mg/kg
  Arms: 1

SUMMARY:
To evaluate the safety and tolerability of a single IV dose of MEDI-557.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of a single IV dose of MEDI-557 administered to healthy adult subjects in 4 dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 45 years at the time of study entry;
* Weight ≤ 90 kg;
* Healthy by medical history and physical examination;
* Normotensive (systolic blood pressure [BP] < 150 mmHg and diastolic BP <90 mmHg);
* Normal electrocardiogram (ECG) at screening (must occur within 21 days before entry into the study);
* Normal spirometry at screening (must occur within 21 days before entry into the study). Normal spirometry is defined as FEV1 (forced expiratory volume in 1 second) and FVC (forced vital capacity) ≥ 80% predicted and an FEV1/FVC > 70%.
* Written informed consent obtained from the subject;
* Sexually active females, unless surgically sterile, must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, abstinence, use of a condom with spermicide by the sexual partner or sterile sexual partner) for 14 days prior to study drug dosing, must agree to continue using such precautions for 1 year after administration of study drug, and must have a negative serum pregnancy test within 3 days prior to study drug dosing and a negative urine pregnancy test on the day of study drug administration; and
* Ability to complete follow-up period of 240 days as required by the protocol.

Exclusion Criteria:

* Acute illness at study entry;
* Fever ≥ 99.5°F at study entry;
* Any drug therapy within 7 days prior to Study Day 0 (except contraceptives);
* Blood donation in excess of 400 mL within 6 months prior to study entry;
* Receipt of immunoglobulin or blood products within 60 days prior to study entry;
* Receipt of any investigational drug therapy or standard vaccine within 120 days prior to study drug dosing through 240 days after study drug dosing;
* Previous receipt of palivizumab or motavizumab; History of immunodeficiency;
* History of allergic disease or reactions likely to be exacerbated by any component of either study drug;
* Previous medical history or evidence of an intercurrent illness that may compromise the safety of the subject in the study;
* Evidence of any systemic disease on physical examination;
* Evidence of infection (ie, positive laboratory test result) with hepatitis A, B, or C virus or human immunodeficiency virus-1 (HIV-1);
* At screening (must be within 21 days before entry into the study) any of the following: hemoglobin < 12.0 gm/dL, white blood cell count (WBC) < 4,000/mm3, platelet count < 120,000/mm3 (or laboratory normal values); aspartate aminotransferase (AST), alanine aminotransferase (ALT), blood urea nitrogen (BUN), serum creatinine > upper limit of normal (ULN); other abnormal laboratory values in the screening panel which, in the opinion of the principal investigator, are judged to be clinically significant; other abnormal laboratory values in the screening panel which, in the opinion of the principal investigator, are judged to potentially confound analysis of study results;
* Pregnancy, or nursing mother;
* History of alcohol or drug abuse within the past 2 years; or
* History of asthma, seasonal allergies, or exercise-induced wheezing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-12; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The occurrence of AEs from the period immediately following study drug administration | through 28 days after dosing
The occurrence of laboratory AEs from the period immediately following study drug administration | through 90 days after dosing
The occurrence of SAEs from the period immediately following study drug administration | through 240 days after dosing

SECONDARY OUTCOMES:
The single-dose pharmacokinetic parameters of IV MEDI-557 and motavizumab monitored using noncompartmental analysis. | Day 240

CONTACTS AND LOCATIONS:
Overall Officials: M. Pamela Griffin, M.D., Study Director — MedImmune LLC
Locations (1):
- Covance Daytona Beach, Daytona Beach, Florida, United States

REFERENCES:
- [Derived] Robbie GJ, Criste R, Dall'acqua WF, Jensen K, Patel NK, Losonsky GA, Griffin MP. A novel investigational Fc-modified humanized monoclonal antibody, motavizumab-YTE, has an extended half-life in healthy adults. Antimicrob Agents Chemother. 2013 Dec;57(12):6147-53. doi: 10.1128/AAC.01285-13. Epub 2013 Sep 30. PMID 24080653